CLINICAL TRIAL: NCT02795403
Title: Hepatitis C Virus Particles-bound Human Proteins : Identification in Clinical Samples and Implication in the Viral Life Cycle
Brief Title: HCV Virions Bound Proteins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2009-596
Record Dates: First submitted 2016-05-17; First posted 2016-06-10 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hepatitis C
Keywords: HCV, liver
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Viraemic (Experimental)
  Interventions: Other: blood draw of 150ml, twice
- responder group (Experimental)
  Interventions: Other: blood draw of 150ml, twice

INTERVENTIONS:
Other: blood draw of 150ml, twice

SUMMARY:
The emergence of hepatocellular carcinoma (HCC) has prompted a search for a thorough understanding of the biology of one of its major causative agents, the hepatitis C virus (HCV). HCV particles acquire via budding and encapsidation cellular proteins. There is mounting evidence on several viral species that virion-bound proteins are prone to be involved either at the replication, budding/egress or entry/release steps of the viral cycle.

Identifying such targets may yield ideal candidates for gaining insight on the dependence of HCV upon a restricted subset of host proteins, therefore providing refined sets of genetically stable targets for therapy. This project's goals are to set up adequate conditions for robust and reproducible purification of HCV virions in clinical samples, followed by the identification of their HCV-bound host proteins and the characterization of their functions. Proteomics profiling of HCV particles purified from clinical samples will be overlaid with proteins identified and characterized in cell culture grown HCV particles during my post-doctoral training, using clinical biomarker discovery grade criteria. Targets identified in both samples sets will be subjected to in vitro investigations using HCV-replicating cells. Conventional biochemical and imaging methods will be used in order to: (i) ascertain their physical association with HCV virions; (ii) define the modalities of their interaction with HCV proteins; (iii) decipher the topology and subcellular localization of their association with HCV proteins and virions; (iv) quantitatively assess their functional involvement in particle budding, egress or secretion and infectivity. A candidate that yielded satisfactory results in these experiments will be disclosed and further investigated at the level of structural biology, in collaborative research programs.

ELIGIBILITY:
Inclusion Criteria:

* Adult> 18 and <60 years
* Infected with HCV genotype 1 HCV antibody positive.
* positive viremia for more than 6 months
* Viremia> 106 IU / ml.
* nonresponders to previous treatment and without antiviral treatment for 2 months.
* For control samples: Patients responders to previous treatment and without antiviral treatment for 2 months.

Exclusion Criteria:

* Patient receiving or having received antiviral treatment within two months.
* patient with against-indication for a blood sample of 150 ml
* immunosuppressive therapy patient
* Patient with liver disease other than hepatitis C.
* Patients with cirrhosis.
* patient with hepatocellular carcinoma.
* Patients with one or more severe co-morbidities defined as:
* Co-infection with HIV or HBV.
* hematological malignancies changing or aplasia
* Insulin-dependent diabetes
* dialyzed chronic renal failure
* Heart failure
* Persons subject to legal protection or the subject of a safeguard measure of justice not affiliated with a social security scheme or not beneficiaries of such a scheme
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Qualitative identification (unit used: Protein Prophet score) of a given virion-bound protein in purified virions preparations | One to two years after mass spectrometry identification of the candidate
  Protein prophet scores allow one to estimate the robustness of identification of a given protein in MS approaches.
Quantitative evaluation of its implication in viral morphogenesis (unit used: TCID50). | One to two years after mass spectrometry identification of the candidate
  TCID50 units are infectivity units routinely used in HCV research for viral infectivity quantification.
Quantitative evaluation of viral entry (unit used: HCV RNA /GUS mRNA copy ratios). | One to two years after mass spectrometry identification of the candidate
  HCV RNA /GUS mRNA copy ratios are derived from the 2^delta(delta Ct) method.

SECONDARY OUTCOMES:
Comparison of clinical virions datasets with in vitro grown virions datasets | One to two years after mass spectrometry identification of the candidate
  Proteins identified from viral particles purified from clinical samples will be compared to proteins identified in viral particles from cells of human hepatocarcinoma (Huh7.5) infected with HCV and from which data are published.

CONTACTS AND LOCATIONS:
Overall Officials: Fabien ZOULIM, MD, Principal Investigator — Service d'Hépato-Gastroentérologie Lyon Croix-Rousse Hospices Civils de Lyon
Locations (1):
- Service d'Hépato-Gastroentérologie Lyon Croix-Rousse Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cottarel J, Plissonnier ML, Kullolli M, Pitteri S, Clement S, Millarte V, Si-Ahmed SN, Farhan H, Zoulim F, Parent R. FIG4 is a hepatitis C virus particle-bound protein implicated in virion morphogenesis and infectivity with cholesteryl ester modulation potential. J Gen Virol. 2016 Jan;97(1):69-81. doi: 10.1099/jgv.0.000331. Epub 2015 Oct 29. PMID 26519381